CLINICAL TRIAL: NCT03245255
Title: Noninvasive Real-time Intracardiac Pressure Measurements Using Subharmonic Ultrasound
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R21HL130899 (NIH); R21HL130899 (NIH)
Record Dates: First submitted 2017-08-04; First posted 2017-08-10 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Catheterization; Blood Pressure; Heart Ventricles; Echocardiography; Heart Failure
Keywords: pressure measurements; blood pressure; contrast echocardiography; ventricular pressures; catheterization
MeSH Terms: conditions — Heart Failure | interventions — Sonazoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sonazoid for pressure measurements (Experimental): 48 µl of Sonazoid microbubbles (GE Healthcare, Oslo, Norway) will be co-infused at a rate of 0.024 µl/kg body weight/minute together with a 0.9% sodium chloride solution infused at a rate of at least 2 ml/min.
  Interventions: Drug: Sonazoid

INTERVENTIONS:
Drug: Sonazoid — Whenever a patient undergoes cardiac catheterization, which routinely includes intracardiac pressure monitoring using a pressure catheter, as part of their standard clinical care and agrees to participate in the study, we will acquire research data. With Sonazoid infusion, SHAPE algorithm will be initiated to determine optimum acoustic pressure. Then, at the optimum acoustic pressure, SHAPE specific data will be acquired from the cardiac chambers and aorta synchronously with the pressures recorded by the catheter (as a part of the patient's standard of care). After acquiring the ultrasound imaging data, the remainder of the heart catheterization will be completed by the attending cardiologist according to the patients' standard of care.

SUMMARY:
This study will use contrast echocardiography to assess the accuracy of a new non-invasive imaging method for subharmonic aided pressure estimation (SHAPE) compared to simultaneously acquired intra-cardiac pressures measured invasively during cardiac catheterization. This study is designed to verify that contrast echocardiography using the SHAPE method, already proven in a canine model and tested in a human pilot study can be used as a surrogate for cardiac catheterization with sufficient accuracy to allow clinical applicability in humans.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for cardiac catheterization procedure.
* Be at least 18 years of age.
* Be medically stable.
* If a female of child-bearing potential, must have a negative pregnancy test.
* Be conscious and able to comply with study procedures.
* Have signed Informed Consent to participate in the study.

Exclusion Criteria:

* Clinically unstable patients, e.g., those who are clinically in decompensated heart failure or having active chest pain or presenting for admission with an unstable anginal syndrome
* Patients in whom introduction of a catheter into the left ventricle is contraindicated or would potentially be dangerous, e.g., patients with active ventricular arrhythmias or with significant aortic valve stenosis where crossing the aortic valve may be difficult and not clinically necessary
* Females who are pregnant or nursing.
* Patients not scheduled for cardiac catheterization procedure.
* Patients who have received an investigational drug in the 30 days before, or will receive one within 72 h after, study drug administration.
* Patients currently on chemotherapy or with other primary cancers requiring treatment.
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable.
* Patients with a history of anaphylactic allergy to eggs or egg products, manifested by one or more of the following symptoms: generalised urticaria, difficulty in breathing, swelling of the mouth and throat, hypotension, or shock. (Subjects with nonanaphylactic allergies to eggs or egg products may be enrolled in the study, but must be watched carefully for 1 h following the administration of SONAZOID).
* Patients with congenital heart defects.
* Patients with severe emphysema, pulmonary vasculitis, or a history of pulmonary emboli.
* Patients with respiratory distress syndrome or a contraindication to pharmacological vasodilator stress agents.
* Patients with thrombosis within the hepatic, portal, or mesenteric veins.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaydev K Dave, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University and Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will generate pressure values in the aorta, and left and right ventricles using the proposed research method (i.e., SHAPE) and using the standard of care (i.e., catheter based pressure values). Additionally peripheral and central pressures will be generated. All of the pressure values will be made available. Further, all ultrasound data obtained for SHAPE measurements will be made available after anonymizing the data-set to remove any patient information
Supporting Information: CSR
Time Frame: 2018-08-01 (anticipated) or starting 6 months after publication
Access Criteria: Accessible research platform

REFERENCES:
- [Background] Dave JK, Halldorsdottir VG, Eisenbrey JR, Liu JB, McDonald ME, Dickie K, Leung C, Forsberg F. Noninvasive estimation of dynamic pressures in vitro and in vivo using the subharmonic response from microbubbles. IEEE Trans Ultrason Ferroelectr Freq Control. 2011 Oct;58(10):2056-66. doi: 10.1109/TUFFC.2011.2056. PMID 21989870
- [Background] Dave JK, Halldorsdottir VG, Eisenbrey JR, Forsberg F. Processing of subharmonic signals from ultrasound contrast agents to determine ambient pressures. Ultrason Imaging. 2012 Apr;34(2):81-92. doi: 10.1177/016173461203400202. PMID 22724314
- [Background] Dave JK, Halldorsdottir VG, Eisenbrey JR, Merton DA, Liu JB, Machado P, Zhao H, Park S, Dianis S, Chalek CL, Thomenius KE, Brown DB, Forsberg F. On the implementation of an automated acoustic output optimization algorithm for subharmonic aided pressure estimation. Ultrasonics. 2013 Apr;53(4):880-8. doi: 10.1016/j.ultras.2012.12.010. Epub 2013 Jan 2. PMID 23347593
- [Background] Dave JK, Halldorsdottir VG, Eisenbrey JR, Raichlen JS, Liu JB, McDonald ME, Dickie K, Wang S, Leung C, Forsberg F. Subharmonic microbubble emissions for noninvasively tracking right ventricular pressures. Am J Physiol Heart Circ Physiol. 2012 Jul;303(1):H126-32. doi: 10.1152/ajpheart.00560.2011. Epub 2012 May 4. PMID 22561300
- [Background] Dave JK, Halldorsdottir VG, Eisenbrey JR, Raichlen JS, Liu JB, McDonald ME, Dickie K, Wang S, Leung C, Forsberg F. Noninvasive LV pressure estimation using subharmonic emissions from microbubbles. JACC Cardiovasc Imaging. 2012 Jan;5(1):87-92. doi: 10.1016/j.jcmg.2011.08.017. PMID 22239898
- [Background] Eisenbrey JR, Dave JK, Halldorsdottir VG, Merton DA, Miller C, Gonzalez JM, Machado P, Park S, Dianis S, Chalek CL, Kim CE, Baliff JP, Thomenius KE, Brown DB, Navarro V, Forsberg F. Chronic liver disease: noninvasive subharmonic aided pressure estimation of hepatic venous pressure gradient. Radiology. 2013 Aug;268(2):581-8. doi: 10.1148/radiol.13121769. Epub 2013 Mar 22. PMID 23525208
- [Background] Forsberg F, Liu JB, Shi WT, Furuse J, Shimizu M, Goldberg BB. In vivo pressure estimation using subharmonic contrast microbubble signals: proof of concept. IEEE Trans Ultrason Ferroelectr Freq Control. 2005 Apr;52(4):581-3. doi: 10.1109/tuffc.2005.1428040. PMID 16060506
- [Background] Halldorsdottir VG, Dave JK, Leodore LM, Eisenbrey JR, Park S, Hall AL, Thomenius K, Forsberg F. Subharmonic contrast microbubble signals for noninvasive pressure estimation under static and dynamic flow conditions. Ultrason Imaging. 2011 Jul;33(3):153-64. doi: 10.1177/016173461103300301. PMID 21842580
- [Background] Shi WT, Forsberg F, Raichlen JS, Needleman L, Goldberg BB. Pressure dependence of subharmonic signals from contrast microbubbles. Ultrasound Med Biol. 1999 Feb;25(2):275-83. doi: 10.1016/s0301-5629(98)00163-x. PMID 10320317
- [Background] Halldorsdottir VG, Dave JK, Eisenbrey JR, Machado P, Zhao H, Liu JB, Merton DA, Forsberg F. Subharmonic aided pressure estimation for monitoring interstitial fluid pressure in tumours--in vitro and in vivo proof of concept. Ultrasonics. 2014 Sep;54(7):1938-44. doi: 10.1016/j.ultras.2014.04.022. Epub 2014 May 6. PMID 24856899
- [Derived] Esposito C, Machado P, McDonald ME, Savage MP, Fischman D, Mehrotra P, Cohen IS, Ruggiero N 2nd, Walinsky P, Vishnevsky A, Dickie K, Davis M, Forsberg F, Dave JK. Evaluation of Intracardiac Pressures Using Subharmonic-aided Pressure Estimation with Sonazoid Microbubbles. Radiol Cardiothorac Imaging. 2024 Feb;6(1):e230153. doi: 10.1148/ryct.230153. PMID 38358329
- [Derived] Esposito C, Machado P, Cohen IS, Mehrotra P, Savage M, Fischman D, Davis M, Ruggiero N, Walinsky P, McDonald ME, Dickie K, Forsberg F, Dave JK. Comparing Central Aortic Pressures Obtained Using a SphygmoCor Device to Pressures Obtained Using a Pressure Catheter. Am J Hypertens. 2022 May 10;35(5):397-406. doi: 10.1093/ajh/hpac010. PMID 35079778

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sonazoid for Pressure Measurements
Started | 80
Completed | 71
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Sonazoid for Pressure Measurements
Number analyzed (Participants) | 80
Age, Continuous [Mean (Full Range); unit: years] | 63 [32 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non Hispanic | 61
  Black or African American | 15
  Asian | 2
  Hispanic or Latino | 1
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 80
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 30 [15 to 49]

OUTCOME MEASURES:

1. Primary Outcome: Agreement Between SHAPE and Pressure Catheter Measurements
Description: The Pearson correlation coefficient was computed between the simultaneously acquired subharmonic signal and pressure catheter data (i.e., waveforms) for each participant. The Pearson correlation coefficient was used for comparing waveforms given the underlying data and pressure values used for comparisons followed a normal distribution. Values reported will be the mean Pearson correlation coefficient values between the subharmonic waveforms and pressure catheter waveforms obtained.
Time Frame: up to 1 day
Population: Data was not acquired in all the enrolled patients due to health concerns during the catheterization procedure, software and/or hardware issues related to the data acquisition process, patient scheduling and/or arrival of emergency cases, and withdrawn consent before the procedure.
Measure: Mean (Standard Deviation); unit: Correlation coefficient value
Groups:
- For Data From Right Ventricle: For cases in which data was acquired from right ventricle
- For Data From Left Ventricle: For cases in which data was acquired from left ventricle
Arm/Group | For Data From Right Ventricle | For Data From Left Ventricle
Number analyzed (Participants) | 22 | 25
Correlation coefficient value | -0.8 (0.1) | -0.8 (0.1)
Statistical Analysis 1: Comparison: For Data From Right Ventricle vs For Data From Left Ventricle; Test type: Other — Correlation analysis; Pearson Correlation Coefficient = -0.8, Standard Deviation 0.1

2. Primary Outcome: Error Between SHAPE and Pressure Catheter Measurements
Description: Based on the distribution of the differences in cardiac pressure values obtained using the SHAPE technique and the clinical pressure catheter, either a two-tailed paired t test (normal distribution) or Wilcoxon signed rank test (nonnormal distribution) was used to compare the SHAPE technique to the reference standard. Bonferroni corrections were used for multiple comparisons
Time Frame: up to 1 day
Population: LV data were acquired in 25 participants; error calculations were not performed in seven (of 25) participants because the subharmonic signal range was less than the noise threshold of 2.5 dB. RV data were acquired in 22 participants. From this set of 22 participants, the aortic data were not acquired in most, as the participants were scheduled for right heart catheterization only. Due to this, we could only process data from the participants with aortic pressure measurements available.
Measure: Median (Standard Deviation); unit: mmHg
Groups:
- For Data From Left Ventricle - Errors in Mean Diastolic Pressure: Errors in mean diastolic pressures between pressures obtained using the pressure catheter and using the SHAPE technique
- For Data From Left Ventricle - Errors in Minimum Diastolic Pressure: Errors in minimum diastolic pressures between pressures obtained using the pressure catheter and using the SHAPE technique
- For Data From Left Ventricle - Errors in End Diastolic Pressure: Errors in end diastolic pressures between pressures obtained using the pressure catheter and using the SHAPE technique
- For Data From Right Ventricle: Errors in systolic pressures between pressures obtained using the pressure catheter and using the SHAPE technique
Arm/Group | For Data From Left Ventricle - Errors in Mean Diastolic Pressure | For Data From Left Ventricle - Errors in Minimum Diastolic Pressure | For Data From Left Ventricle - Errors in End Diastolic Pressure | For Data From Right Ventricle
Number analyzed (Participants) | 18 | 18 | 18 | 8
mmHg | 5.4 (7.4) | 6.6 (8.3) | 5.8 (7.5) | 1.2 (1.5)

ADVERSE EVENTS:
Time Frame: During data acquisition after Sonazoid infusion (5-10 minutes) and when the patients were observed in the recovery area after the procedure for up to 60 minutes after the procedure.
Arm/Group | Sonazoid for Pressure Measurements
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT03245255/Prot_SAP_000.pdf